CLINICAL TRIAL: NCT04186364
Title: Implementation and Evaluation of the Autism Spectrum Ambassador Program
Brief Title: Autism Spectrum Ambassador Program (ASAP) in the ED
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to COVID-19 pandemic.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Cheryl Tierney, Associate Professor of Pediatrics, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00002020
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Austism; Ambassador
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assigned Ambassador (Intervention Group) (Experimental): Patients who were consented, completed the accommodations survey, and for whom a medical student was available during the time of the ED visit will serve as our intervention group. The participants will be assigned an Ambassador throughout the child's ED visit and will complete a patient satisfaction survey afterwards. The investigators hold to enroll 120 controls.
  Interventions: Behavioral: Assigned Ambassador
- Control Group (No Intervention): Patients who were consented, completed the accommodations survey, but for whom a medical student was not available during the time of the ED visit will serve as our control group. The controls will fill out both an accommodations survey before and a patient satisfaction survey after the ED visit, however no ambassador will be assigned during the ED visit. The investigators hope to enroll 120 controls.

INTERVENTIONS:
Behavioral: Assigned Ambassador — If assigned to the intervention group, participants will be assigned a medical student ambassador on arrival to the Emergency Department. A brief discussion may take place to review the child's history and survey results, and a copy of the survey will be placed near the patient's bedside for healthcare personnel to review. The student ambassador will accompany the child and their family through key points of their visit and will be expected to make accommodations for the child as determined by the accommodation survey results. The family will be required to allow the ambassador to stay throughout the ED visit.
  Arms: Assigned Ambassador (Intervention Group)

SUMMARY:
The investigators are evaluating the implementation and the effectiveness of a medical student staffed support program (ASAP) for children diagnosed with Autism Spectrum Disorder coming into Penn State Hershey Children's Hospital Emergency Department. The ASAP program involves training and assigning a medical student as an Ambassador to help advocate for the special needs of a child with ASD. This study is designed to compare patient satisfaction of children and families who are assigned an Ambassador to those who are not assigned an Ambassador during their time in the Emergency Department. The secondary objectives are to measure overall medical student satisfaction with the program, medical student career interests before and after participation, and medical student comfort level interacting with children with ASD before and after participation.

DETAILED DESCRIPTION:
The Autism Spectrum Ambassador Program (ASAP) is a medical student staffed program designed to improve the experience for children with Autism Spectrum Disorder coming into the Children's Hospital Emergency Department (ED) for an acute visit. This program will pair an interested and trained medical student with a family whose child presents to the Children's Hospital ED and identifies as having Autism and requiring special accommodations to improve cooperation and procedure tolerance.

Patients will be identified by the study team members, who are ages 30 months to 17years with the diagnosis of Autism Spectrum Disorder. Participants will be recruited through posters and flyers in the Pediatric Emergency Room Waiting area; families who are interested in enrolling will enter the research study. Interested caregivers will be asked to complete a confidential survey that will identify areas that can be accommodated during their visit. This survey will then be automatically be printed for the ED staff and ambassador to review. The student will meet the family in the ED and accompany the family through their visit; the student will print the child's Accommodation Plan, place it at the bedside, and make it available for each member of the treatment team.

Students will be trained to chart a child's Accommodation Plan for each member of the treatment team and place it at bedside, as well to advocate on behalf of the child and their family, communicate with the staff (including nurses, primary care providers (physicians and Physician Assistants (PAs)), and techs (radiology, phlebotomy, transport). To the extent possible, the investigators hope that having a student advocate, educate staff in the ED, and implement changes as needed will improve patient satisfaction with the experience and improve the ease with which a procedure can be carried out for a child with ASD. Students will also be queried as to the experience and survey data will be used to improve the program over time.

Training will be completed so that all members of the treatment team will be aware of the program and aware of the possible accommodations. Treatment team members will be provided additional training to enhance the success of the ASAP program and all treatment team members will be encouraged to work together for the best possible outcome for all patients. Treatment team services include: nursing, ED physicians, PAs, technicians (radiology, phlebotomy, transport), registration, and to the extent possible, the personnel involved in the care of these children.

ELIGIBILITY:
Inclusion Criteria:

1. Study Participants:

1. Must be children 30 months to 17 years of age.
2. Study participants will be boys and girls.
3. Study participants will have a a diagnosis of Autism Spectrum Disorder.
4. Study participants will be presenting through the pediatric emergency room at the Penn State Hershey Medical Center.
5. Study participants must be English Speaking.

2. Medical Student Ambassadors:

1. Ambassadors must be enrolled as first, second, third, or fourth year medical students at the Penn State College of Medicine
2. Ambassadors must complete training successfully

Exclusion Criteria:

1. Study Participants:

1. Children under 30 months or older than 17 years.
2. Children who do not have a diagnosis of Autism Spectrum Disorder.
3. Children who cannot understand and communicate in English.

2. Medical Student Ambassadors:

1. Individuals who are not a medical student at the Penn State College of Medicine.
2. Medical students who do not complete the training course.
3. Medical students who are not deemed appropriate the ASAP Ambassador role as per the discretion of study personnel.

Ages: 30 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction Survey (Questionnaire) | 1 year.
  Improved patient satisfaction and fewer behavioral complications during the procedure day; data collected using REDCap. The questionnaire, likely titled "ASAP Patient Satisfaction Survey", will include scales of 0-10 rating satisfaction in various categories with 10 being extremely satisfied and 0 being very unsatisfied.

SECONDARY OUTCOMES:
Medical Student Satisfaction Survey (Questionnaire) | 1 year
  Overall medical student satisfaction with the ambassador program; data collected using REDCap.The questionnaire, likely titled "ASAP Medical Student Satisfaction Survey", will include scales of 0-10 rating satisfaction in various categories with 10 being extremely satisfied and 0 being very unsatisfied.
Medical Student Career Interest (Questionnaire) | 1 year
  Medical student career interests before and after participation in this program; data collected using REDCAP. The questionnaire, likely titled "Impact of ASAP on Career Interest" may include scales of 0-10 rating satisfaction in various categories with 10 being extremely satisfied and 0 being very unsatisfied but will also include unscaled questions with answers such as "very interested, somewhat interested, not interested, etc.".
Medical Student Comfort Level (Questionnaire) | 1 year
  Medical student comfort level interacting with autistic children before and after participation in the program; data collected using REDCap.The questionnaire, likely titled "Impact of ASAP on Medical Student Comfort Levels with Patients with Autism", may include scales of 0-10 rating satisfaction in various categories with 10 being extremely satisfied and 0 being very unsatisfied among unscaled questions with answers such as "very comfortable, neutral, and very uncomfortable."

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Tierney, M.D., Principal Investigator — Developmental Pediatrics, Penn State Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Gimbler Berglund I, Huus K, Enskar K, Faresjo M, Bjorkman B. Perioperative and Anesthesia Guidelines for Children with Autism: A Nationwide Survey from Sweden. J Dev Behav Pediatr. 2016 Jul-Aug;37(6):457-64. doi: 10.1097/DBP.0000000000000289. PMID 27011004
- [Background] Nayfack AM, Huffman LC, Feldman HM, Chan J, Saynina O, Wise PH. Hospitalizations of children with autism increased from 1999 to 2009. J Autism Dev Disord. 2014 May;44(5):1087-94. doi: 10.1007/s10803-013-1965-x. PMID 24122446
- [Background] Broder-Fingert S, Shui A, Ferrone C, Iannuzzi D, Cheng ER, Giauque A, Connors S, McDougle CJ, Donelan K, Neumeyer A, Kuhlthau K. A Pilot Study of Autism-Specific Care Plans During Hospital Admission. Pediatrics. 2016 Feb;137 Suppl 2:S196-204. doi: 10.1542/peds.2015-2851R. PMID 26908475
- See also: Study Protocol — http://irb.psu.edu
- See also: Informed Consent Form — http://irb.psu.edu
- See also: Accommodation Survey — http://irb.psu.edu
- See also: Patient Satisfaction Survey — http://irb.psu.edu
- See also: Medical Student Survey — http://irb.psu.edu
- See also: Summary Explanation of Research - for Medical Students — http://irb.psu.edu